CLINICAL TRIAL: NCT02864082
Title: A Randomized, Bilateral Comparison, Vehicle-Controlled, Safety and Tolerability Study of Topical PAT-001 for the Treatment of Congenital Ichthyosis
Brief Title: A Safety and Tolerability Study of Topical PAT-001 in Congenital Ichthyosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patagonia Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205-9051-201
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Congenital Ichthyosis
Keywords: X-linked, lamellar
MeSH Terms: conditions — Ichthyosis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PAT-001 0.1% (Experimental): Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.1% (e.g., left side) and Vehicle, 0.0% (e.g., right side). This comparison lasts from Weeks 0-8 Part 2: Patients will apply only PAT-001, 0.1% to both Treatment Areas from Weeks 8-12.
  Interventions: Drug: PAT-001, 0.1%
- PAT-001 0.2% (Experimental): Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.2% (e.g., left side) and Vehicle, 0.0% (e.g., right side). This comparison lasts from Weeks 0-8 Part 2: Patients will apply PAT-001, 0.2% to both Treatment Areas.
  Interventions: Drug: PAT-001, 0.2%
- Vehicle for PAT-001 0.1% arm (Placebo Comparator): Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.1% (e.g., left side) and Vehicle, 0.0% (e.g., right side). The application of vehicle only lasts from Weeks 0-8.
  Interventions: Drug: Vehicle for PAT-001 0.1%
- Vehicle for PAT-001 0.2% arm (Placebo Comparator): Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.2% (e.g., left side) and Vehicle, 0.0% (e.g., right side). The application of vehicle only lasts from Weeks 0-8.
  Interventions: Drug: Vehicle for PAT-001 0.2%

INTERVENTIONS:
Drug: PAT-001, 0.1% — PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
  Other Names: PAT-001
  Arms: PAT-001 0.1%
Drug: PAT-001, 0.2% — PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
  Other Names: PAT-001
  Arms: PAT-001 0.2%
Drug: Vehicle for PAT-001 0.1% — Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001 0.1%.
  Other Names: Vehicle
  Arms: Vehicle for PAT-001 0.1% arm
Drug: Vehicle for PAT-001 0.2% — Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001 0.2%.
  Other Names: Vehicle
  Arms: Vehicle for PAT-001 0.2% arm

SUMMARY:
Congenital ichthyosis (CI) is a large, heterogeneous family of inherited skin disorders of cornification resulting from an abnormality of skin keratinization, such as scaling and thickening of the skin. Treatment options include keratolytic agents, which can abruptly lead to extensive shedding or peeling of scales. PAT-001 primarily acts as a keratolytic agent; thus, making it a potential drug candidate for the treatment of skin disorders associated with hyperkeratinization, such as CI. The current study intends to evaluate the safety and tolerability of PAT-001 in patients with CI of either the Lamellar or X-Linked subtypes.

DETAILED DESCRIPTION:
The management of CI is a life-long endeavor, which remains largely symptomatic (i.e., emollients with or without keratolytics agents) and commonly focused on reducing scaling and/or skin lubrication with both systemic and topical treatments. A first-line therapy includes hydration and lubrication accomplished by creams and ointments containing low concentrations of salt, urea, or glycerol, which increase the water-binding capacity of the horny layer. Addition of keratolytics agents are used to decrease corneocyte cohesiveness, to promote desquamation, and to dissolve keratins and lipids (e.g., α-hydroxy acids, salicylic acid, high dose urea, propylene glycol, N-acetylcysteine, and retinoids). Systemic retinoid treatment is reserved for those patients refractory to topical agents because of long-term adverse effects and teratogenicity.

This is a two part, Phase 2, multicenter, proof-of-concept (POC) study of the safety and tolerability of PAT-001 for the treatment of Congenital ichthyosis (CI) in patients ages 12 years of age and older. Part 1 will be a double-blind, randomized, vehicle controlled, bilateral comparison of two treatments (PAT-001 [0.1% or 0.2%] vs. vehicle) for eight (8) weeks.

Part 2 will be a double-blind, active only treatment comparison of the two PAT-001 concentrations (0.1% or 0.2%) for an additional four (4) weeks. Subjects will have the option to participate in the pharmacokinetics (PK) portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 12 years or older.
* Females of childbearing potential should use appropriate contraception. Women of childbearing potential must have a negative pregnancy test at screening and baseline visits.
* Patient and legal representative(s), if applicable, has provided written informed consent.
* Patient has congenital ichthyosis of either lamellar or X-Linked subtype.
* Patient has two contralateral comparable Treatment Areas (e.g., each arm is affected and treatments areas can be applied equally).
* Patient is, except for their ichthyosis, in good general health.

Exclusion Criteria:

* Patient is pregnant or breast feeding, or is planning to become pregnant during the study.
* Patient has inflammatory skin disease unrelated to ichthyosis.
* Patient is currently using concomitant retinoid therapy, within two weeks (topical) or 12 weeks (oral) of Visit 2/Baseline.
* Patient is currently taking concomitant immunosuppressive drugs, including systemic corticosteroids, within two weeks of Visit 2/Baseline.
* Patient is currently enrolled in an investigational drug or device study.
* Patient has used an investigational drug or investigational device treatment within 30 days prior to Visit 2/Baseline.
* Patient is unable to communicate or cooperate with the investigator due to language problems, impaired cerebral function, or physical limitations.
* Patient is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Rome, BS, Study Director — Sponsor GmbH
Locations (5):
- United States (5):
  - TCR Medical Corporation, San Diego, California
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Paddington Testing Co., Inc, Philadelphia, Pennsylvania
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: March 8, 2017-February 13, 2018. Recruited at 5 clinics in United States associated with US Universities by practicing dermatologists
Pre-assignment Details: Each patient received both vehicle application and either PAT-001 0.1% or PAT-001 0.2% on 2 different identical matching parts of their bodies (e.g, upper thighs). Since each of the 19 patients were treated with both PAT-001 and vehicle, the number of treatment areas was 38 (19 x 2) but the number of patients was 19.
Groups:
- Group 1 PAT-001 0.1% and Vehicle: Part 1 (8 weeks): Patients will have two comparable Treatment Areas on their bodies, for example both upper arms that have same degree of disease. PAT-001, 0.1% will be applied to one of those body parts for 8 weeks, applied twice a day. The matching body part will have vehicle applied twice a day for 8 weeks
  Part 2 (4 weeks): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001 0.1% so that subjects cannot tell the difference between vehicle and PAT-001 based upon appearance.
- Group 2 PAT-001 0.2% and Vehicle: Part 1 (8 weeks): Patients will have two comparable Treatment Areas on their bodies, for example both upper arms that have same degree of disease. PAT-001, 0.2% will be applied to one of those body parts for 8 weeks, applied twice a day. The matching body part will have vehicle applied twice a day for 8 weeks.
  Part 2 (4 weeks): Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001 0.1% so that subjects cannot tell the difference between vehicle and PAT-001 based upon appearance.
Period: Overall Study
Arm/Group | Group 1 PAT-001 0.1% and Vehicle | Group 2 PAT-001 0.2% and Vehicle
Started | 10 | 9
Completed | 7 | 5
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1 PAT-001 0.1% and Vehicle: Part 1 (weeks 0-8): Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.1% (e.g., left side) and Vehicle, 0.0% (e.g., right side).
  Part 2 (weeks 8-12): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
- Group 2 PAT-001 0.2% and Vehicle: Part 1 (weeks 0-8): Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.2% (e.g., left side) and Vehicle, 0.0% (e.g., right side).
  Part 2: (weeks 8-12) Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
- Total: Total of all reporting groups
Arm/Group | Group 1 PAT-001 0.1% and Vehicle | Group 2 PAT-001 0.2% and Vehicle | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (20.3) | 47.2 (18.4) | 42 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28.8 [19 to 33.9] | 26.4 [18 to 41.2] | 27.7 [18 to 41.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) in Part 1 of Trial (Weeks 0-8)
Description: The number of participants with AEs will be assessed by the investigator and the incidence (severity and causality) of any local and systemic AEs will be reported.
Time Frame: Day 0 through Day 57 (Weeks 0-8)
Population: Number of Participants with Adverse events
Measure: Number; unit: participants
Groups:
- Group 1 PAT-001 0.1%: Part 1 (Weeks 0-8): Patients will have two comparable Treatment Areas of equal size and degree of severity: PAT-001, 0.1% will be applied to one of the 2 areas twice a day for 8 weeks
  Part 2 (Weeks 8-12): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
- Group 2 PAT-001 0.2%: Part 1 (Weeks 0-8): Patients will have two comparable Treatment Areas of equal size and degree of severity: PAT-001, 0.2% will be applied to one of the 2 areas twice a day for 8 weeks
  Part 2 (weeks 8-12): Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
- Group 1 Vehicle; Group 2 Vehicle: Part 1 (Weeks 0-8): Patients will have two comparable Treatment Areas of equal size and degree of severity: Vehicle will be applied to one of the 2 areas twice a day for 8 weeks
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
Arm/Group | Group 1 PAT-001 0.1% | Group 2 PAT-001 0.2% | Group 1 Vehicle | Group 2 Vehicle
Number analyzed (Participants) | 10 | 9 | 10 | 9
participants
  Number of Subjects with TEAE | 7 | 7 | 5 | 5
  Number of Treatment Emergent Adverse Events (TEAE) within treatment area | 4 | 5 | 3 | 3
  Number of Deaths due to TEAE | 0 | 0 | 0 | 0
  Number of Serious TEAE | 0 | 1 | 0 | 0
  Number of Patients who Discontinued in the trial due to TEAE | 1 | 1 | 0 | 0
  Number of Patients with Severe TEAE | 1 | 1 | 0 | 0
  Number of Patients with Moderate TEAE | 3 | 3 | 2 | 2
  Number of Patients with Mild TEAE | 4 | 6 | 3 | 3
  Number of Patients Where the TEAE was Considered Definitely Related to Treatment | 1 | 1 | 0 | 0
  Number of Patients where the TEAE was Considered Probably Related to Treatment | 1 | 0 | 0 | 0
  Number of Patients Where the TEAE was Considered Possibly Related to Treatment | 1 | 4 | 1 | 1
  Number of Patients Where the TEAE was Considered Not Related to Treatment | 1 | 5 | 4 | 4

2. Primary Outcome: Incidence of Local Skin Reactions (LSRs) in Participants Treated With PAT-001 0.1%, 0.2% and/or Vehicle
Description: LSRs including burning/stinging, pain, and pruritus (itch) will be assessed in each Treatment Area using a four-point ordinal scale where 0=none, 1=mild, 2=moderate, and 3=severe (based on the investigator's evaluation of the skin reaction) at each clinic visit to allow a comparison between Treatment Groups and Test Articles. Only LSRs that require medical intervention (e.g., prescription medication) or require withholding or reduction in dosing frequency of the test articles will be documented in this LSR Table. Any LSRs that are not listed here will be recorded as AEs.
Time Frame: Up to Day 84 (Weeks 0-12)
Population: Participants may have had more than one type of LSR
Measure: Number; unit: participants
Groups:
- Group 1 PAT-001 0.1%: Part 1 (weeks 0-8): Bilateral randomized comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.1% is applied to one side Part 2 (weeks 8-12): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
- Group 1 Vehicle: Part 1 (weeks 0-8): Bilateral randomized comparison. Patients will have two comparable Treatment Areas: Vehicle, 0.0% will be applied to one of the sides Part 2 (weeks 8-12): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
- Group 2 PAT-001 0.2%: Part 1 (weeks 0-8): Bilateral randomized comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.2% will be applied to one side Part 2 (weeks 8-12): Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
- Group 2 Vehicle: Part 1 (weeks 0-8): Bilateral randomized comparison. Patients will have two comparable Treatment Areas: PAT-001 Vehicle, 0.0% will be applied to one side Part 2 (weeks 8-12): Patients will apply PAT-001, 0.2% to both Treatment Areas.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
Arm/Group | Group 1 PAT-001 0.1% | Group 1 Vehicle | Group 2 PAT-001 0.2% | Group 2 Vehicle
Number analyzed (Participants) | 10 | 10 | 9 | 9
participants
  Application site pruritis (severe) | 1 | 0 | 0 | 0
  Application site irritation (mild) | 3 | 2 | 0 | 0
  Application site dermatitis (moderate) | 0 | 0 | 1 | 0
  Application site rash (mild) | 1 | 0 | 0 | 1
  Application site reaction (mild) | 0 | 0 | 1 | 0
  Application site pain (moderate) | 1 | 0 | 0 | 0
  Application site Pruritis (moderate) | 1 | 1 | 0 | 0
  Application site Pruritis (mild) | 1 | 1 | 0 | 0
  Application site Dermatitis (mild) | 0 | 0 | 1 | 2

3. Secondary Outcome: Number of Participants Achieving Improvement to State of Clear, Almost Clear or Mild in the Investigator's Global Assessment (IGA) Using a Five-point Scale at Day 57 (Part 1)
Description: Overall severity of ichthyosis will be graded using a five-point scale Investigator Global Assessment (IGA) based upon a 5 point scale going from 0=clear., 1=almost clear, 2=mild, 3=moderate to 4=severe. Scoring is based upon investigator evaluation. This is a static morphological scale that refers to a point in time and not a comparison to Baseline.
Time Frame: Up to Day 57
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 PAT-001 0.1%; Group 1 Vehicle: Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.1% (e.g., left side) and Vehicle, 0.0% (e.g., right side).
  Part 2: Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
- Group 2 PAT-001 0.2%; Group 2 Vehicle: Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.2% (e.g., left side) and Vehicle, 0.0% (e.g., right side).
  Part 2: Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
Arm/Group | Group 1 PAT-001 0.1% | Group 2 PAT-001 0.2% | Group 1 Vehicle | Group 2 Vehicle
Number analyzed (Participants) | 9 | 8 | 9 | 8
Participants | 9 | 8 | 6 | 7

4. Secondary Outcome: Number of Participants Achieving an Improvement of at Least 1 Point Score in the Individual Clinical Signs/Symptoms of Erythema, Scaling, Fissuring and Papulation/Lichenification Using a Five-point Scale
Description: Overall severity of erythema (redness), scaling , fissuring (cracks in skin), and papulation/lichenification (skin thickening, increased pigmentation and/or exaggerated skin lines, formation of papules) will be graded using a five-point scale from 0=clear, 1=almost clear, 2=mild, 3=moderate to 4=severe. This is a static morphological scale that refers to a point in time and not a comparison to Baseline. This scoring is based upon investigator discretion.
Time Frame: Up to Day 57 (Weeks 0-8)
Population: IGA score improvement of at least 1 point on IGA for scaling, erythema, papulation/lichenification and fissuring at Day 57 in patients receiving continuous 0.1% and 0.2% PAT-001
Measure: Number; unit: participants
Arm/Group | Group 1 PAT-001 0.1% | Group 2 PAT-001 0.2% | Group 1 Vehicle | Group 2 Vehicle
Number analyzed (Participants) | 9 | 8 | 9 | 8
participants
  Scaling | 9 | 6 | 7 | 8
  Fissuring | 6 | 6 | 5 | 6
  Papulation/lichenification | 9 | 6 | 6 | 7
  Erythema | 5 | 5 | 4 | 6

5. Other Pre Specified Outcome: Pharmacokinetics of PAT-001 0.1% and 0.2% at Different Timepoints
Description: Serum concentrations for PAT-001 0.1% and PAT-001 0.2% looking at blood levels obtained at timepoints outlined
Time Frame: Day 1 (0,1, 2, 3, and 4 hours post Dose)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 1: Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.1% (e.g., left side) and Vehicle, 0.0% (e.g., right side).
  Part 2: Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
- Group 2 (Part 1): Part 1: Bilateral comparison. Patients will have two comparable Treatment Areas: PAT-001, 0.2% (e.g., left side) and Vehicle, 0.0% (e.g., right side).
  Part 2: Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
Arm/Group | Group 1 | Group 2 (Part 1)
Number analyzed (Participants) | 2 | 3
ng/mL
  Pre-Dose | 1.495 (0.6718) | 2.48 (1.795)
  1 Hour | 1.5 (0.6505) | 2.227 (1.3725)
  2 Hours | 1.425 (0.5303) | 2.12 (1.2257)
  3 Hours | 1.37 (0.297) | 2.063 (1.5332)
  4 Hours | 1.375 (0.0778) | 1.453 (0.3625)

ADVERSE EVENTS:
Time Frame: 84 Days
Groups:
- Group 1 PAT-001 0.1%: Part 1 (weeks 0-8) Patients will have two comparable identical Treatment Areas: PAT-001, 0.1% will be applied to one of these areas.
  Part 2 (weeks 8-12): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
- Group 2 PAT-001 0.2%: Part 1 (weeks 0-8) Patients will have two comparable identical Treatment Areas: PAT-001, 0.2% will be applied to one of these areas.
  Part 2 (weeks 8-12): Patients will apply PAT-001, 0.2% to both Treatment Areas.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
- Group 1 Vehicle: Part 1 (weeks 0-8) Patients will have two comparable identical Treatment Areas: Vehicle, 0.0% will be applied to one of these areas.
  Part 2 (weeks 8-12): Patients will apply PAT-001, 0.1% to both Treatment Areas.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
  PAT-001, 0.1%: PAT-001 is a topical ointment. PAT-001, 0.1% contains 0.1% of active drug.
- Group 2 Vehicle: Part 1 (weeks 0-8) Patients will have two comparable identical Treatment Areas: Vehicle 0.0% will be applied to one of these areas.
  Part 2 (weeks 8-12): Patients will apply PAT-001, 0.2% to both Treatment Areas.
  Vehicle: Vehicle topical ointment contains 0.0% of active drug and is color matched to the active test article, PAT-001.
  PAT-001, 0.2%: PAT-001 is a topical ointment. PAT-001, 0.2% contains 0.2% of active drug.
Arm/Group | Group 1 PAT-001 0.1% | Group 2 PAT-001 0.2% | Group 1 Vehicle | Group 2 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 7/10 | 7/9 | 2/10 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 PAT-001 0.1% (N=10) | Group 2 PAT-001 0.2% (N=9) | Group 1 Vehicle (N=10) | Group 2 Vehicle (N=9)
C. difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Deemed not related to study treatment
Novavirus gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 PAT-001 0.1% (N=10) | Group 2 PAT-001 0.2% (N=9) | Group 1 Vehicle (N=10) | Group 2 Vehicle (N=9)
Application site pruritis (General disorders) | 3 (6) | 0 (0) | 2 (2) | 1 (1) — skin reactions
C. difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis novovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data should be interpreted with caution due to small sample sizes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT02864082/Prot_SAP_001.pdf